CLINICAL TRIAL: NCT02375763
Title: Dietary Analysis for Caries Prevention in Children Using a Computer Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Matina Angelopoulou, Assistant Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HR-2908
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sortware suggestions (Experimental): Children will fill a questionnaire regarding their dietary habits. Afterwards a dietary analysis will be performed using a computer software, and dietary instructions will be given to the children.
  Interventions: Other: Software instruction
- Traditional suggestions (Placebo Comparator)
  Interventions: Other: Software instruction

INTERVENTIONS:
Other: Software instruction

SUMMARY:
Children will be recruited from the pediatric dentistry clinic of Marquette University at their first or recall appointment and will be asked to fill a questionnaire regarding their dietary habits. Afterwards a dietary analysis will be performed using a computer software, developed for this study and dietary instructions will be given to the children.

ELIGIBILITY:
Inclusion Criteria:

* Free medical history
* Informed Consent

Exclusion Criteria:

* General disease

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in dietary habits at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University Pediatric Dentistry Clinic, Milwaukee, Wisconsin, United States